CLINICAL TRIAL: NCT02082704
Title: Interactive Spaced Education to Optimize Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AHRQ 1R01HS019708-01A1
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
Keywords: Diabetes; Education, Patient; Educational Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SE Game on DSME (Experimental): The intervention cohort will participate in an online team-based game on diabetes self-management education (DSME) and will receive a paper documents on American history,
  Interventions: Behavioral: SE Game on DSME
- SE Game on American History (Active Comparator): The 'attention control' cohort will participate in an online team-based game on American history and will receive a paper documents on DSME.
  Interventions: Behavioral: SE Game on American History

INTERVENTIONS:
Behavioral: SE Game on DSME — Investigators created an online educational game by incorporating game mechanics into an evidence-based form of online education, termed 'spaced education' (SE). Based upon two psychology research findings (the spacing and testing effects), SE has been shown in randomized trials to improves knowledge acquisition, boosts learning retention for up to two years, and durably improves clinical behavior.
  Arms: SE Game on DSME
Behavioral: SE Game on American History — Investigators created an online educational game by incorporating game mechanics into an evidence-based form of online education, termed 'spaced education' (SE). Based upon two psychology research findings (the spacing and testing effects), SE has been shown in randomized trials to improves knowledge acquisition, boosts learning retention for up to two years, and durably improves clinical behavior.
  Arms: SE Game on American History

SUMMARY:
Investigators are conducting a randomized controlled trial to determine whether an online team-based spaced education (SE) game can improve HbA1c levels among these patients with diabetes (primary aim). Secondary aims include determining the impact of the game on patients' pill possession ratio (PPR) of oral DM meds and their microalbumin/creatinine (M/C) ratio, ACE PPR, and ARB PPR.

DETAILED DESCRIPTION:
Participants will be randomized to one of two cohorts: (1) the intervention cohort will participate in an online team-based game on diabetes self-management education (DSME) and will receive a paper documents on American history, and (2) the 'attention control' cohort will participate in an online team-based game on American history and will receive a paper documents on DSME. Each game would consist of 2 questions per week x 25 weeks = 50 questions total per arm. The questions are delivered via email by the Qstream platform to the participants. Upon clicking on a hyperlink in the email, participants select an answer that is downloaded to a server. They are then provided with the answer to and explanation of the question, along with additional educational materials. Using an adaptive methodology, the spacing and content of the game material will be individualized for each clinician based on their performance. Home-based testing of HbA1c and M/C ratio will be conducted by patients at enrollment, 6 months and 12 months. If successful, this SE game will improve diabetes management among VA patients and improve patient outcomes. Given the growing use of email and the Internet by patients, SE games could be easily expanded to a broad audience of VA patients with varying health problems across the country. With content tailored to meet specific needs, SE games can be utilized as tools to improve patients' clinical outcomes by bolstering their health management behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the northeastern Veterans Affairs hospital system who are taking oral diabetes medications, have a PPR<80%, and have a HbA1c >7.5.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | Months 1-12

SECONDARY OUTCOMES:
Microalbumenuria levels [microalbumin-creatinine ratio]. | Months 1-12
Pill possession ratios of oral diabetes medications. | Months 1-12
Treatment with angiotensin receptor blockers (ARB drugs) and angiotensin converting enzyme inhibitors (ACE inhibitors). | Months 1-12
Pill possession ratios of angiotensin receptor blockers (ARB drugs) and angiotensin converting enzyme inhibitors (ACE inhibitors). | Months 1-12
Weight / BMI | Months 1-12
Low-density lipoprotein (LDL), high-density lipoprotein (HDL), total cholesterol & triglyceride levels, | Months 1-12
Systolic and diastolic blood pressure. | Months 1-12
Clinic visit frequency. | Months 1-12
Initiation or alteration of insulin therapy | Months 1-12
Changes in oral diabetes medication regimen. | Months 1-12
Patient-perceived empowerment to manage their diabetes. | Months 1-12
  Questionnaire
Baseline knowledge levels of patients assessed via their initial responses to SE game questions -- DSME SE game cohort only. | Months 1-6
Analysis of SE game performance differences by patient-related variables (age, gender, geographic location, baseline HbA1c, etc.) -- DSME SE game cohort only. | Months 1-6
Patient-perceived acceptability of SE game interventions. | Months 1-6
  Questionnaire
Patient-perceived barriers and facilitators to the SE game intervention. | Months 1-6
  Questionnaire
Patient's perceptions of the optimal parameters for the SE game intervention. | Months 1-6
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: B. Price Kerfoot, MD EdM, Principal Investigator — VA Boston Healthcare System; Paul R. Conlin, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- Veterans Affairs Boston Healthcare System, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kerfoot BP, Gagnon DR, McMahon GT, Orlander JD, Kurgansky KE, Conlin PR. A Team-Based Online Game Improves Blood Glucose Control in Veterans With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Sep;40(9):1218-1225. doi: 10.2337/dc17-0310. Epub 2017 Aug 8. PMID 28790131